CLINICAL TRIAL: NCT00054236
Title: Pilot Study Of Multiple Umbilical Cord Blood Unit Transplantation Following Non-Myeloablative Conditioning In Patients With Hematologic Disorders Or Severe Aplastic Anemia
Brief Title: Combination Chemotherapy Followed By Umbilical Cord Blood Transplantation in Treating Patients With Hematologic Cancer or Severe Aplastic Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU6Y01
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; adult erythroleukemia (M6a); childhood acute erythroleukemia (M6); adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); adult acute megakaryoblastic leukemia (M7); childhood acute megakaryocytic leukemia (M7); adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; previously treated myelodysplastic syndromes; refractory chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent/refractory childhood Hodgkin lymphoma; polycythemia vera; primary myelofibrosis; essential thrombocythemia; refractory multiple myeloma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent mantle cell lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; Burkitt lymphoma; anaplastic large cell lymphoma; recurrent adult Hodgkin lymphoma; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; atypical chronic myeloid leukemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Large-Cell, Anaplastic; Hodgkin Disease; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Antilymphocyte Serum; Filgrastim; Cyclophosphamide; fludarabine phosphate; Cord Blood Stem Cell Transplantation; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non-myeloablative conditioning regimen (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: cyclophosphamide; Drug: fludarabine phosphate; Procedure: umbilical cord blood transplantation; Drug: methylprednisolone

INTERVENTIONS:
Biological: anti-thymocyte globulin — anti-thymocyte globulin (ATG) IV over at least 4 hours on days -2 to -1
Biological: filgrastim — Patients receive filgrastim (G-CSF) subcutaneously beginning on day 7 and continuing until blood counts recover.
Drug: cyclophosphamide — cyclophosphamide IV over 2 hours on days -3 to -2
Drug: fludarabine phosphate — fludarabine IV over 30 minutes on days -8 to -4
Procedure: umbilical cord blood transplantation — Patients undergo multiple unit umbilical cord blood transplantation on days 0-1.
Drug: methylprednisolone — Patients unable to tolerate ATG may receive methylprednisolone IV over 1 hour on days -3 to -1.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Umbilical cord blood transplantation may be able to replace cells destroyed by chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy followed by umbilical cord blood transplantation in treating patients who have hematologic cancer or severe aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence and severity of acute toxicity in patients with hematologic malignancies or severe aplastic anemia treated with a non-myeloablative conditioning regimen followed by umbilical cord blood transplantation.
* Determine the incidence and severity of acute and chronic graft-versus-host-disease in patients treated with this regimen.
* Determine the incidence of relapse, disease-free survival, and overall survival of patients treated with this regimen.
* Determine the survival rate at 100 days post-transplantation in patients treated with this regimen.
* Determine the incidence of regimen-related complications (infection, hepatic veno-occlusive disease, and interstitial pneumonitis) in patients treated with this regimen.
* Determine the incidence of primary and secondary graft failure in patients treated with this regimen.
* Determine the rates and kinetics of donor-derived lymphoid, myeloid, neutrophil, RBC, and platelet engraftment in patients treated with this regimen.

OUTLINE: Patients receive a non-myeloablative conditioning regimen comprising fludarabine IV over 30 minutes on days -8 to -4, cyclophosphamide IV over 2 hours on days -3 to -2, and anti-thymocyte globulin (ATG) IV over at least 4 hours on days -2 to -1. Patients unable to tolerate ATG may receive methylprednisolone IV over 1 hour on days -3 to -1.

Patients undergo multiple unit umbilical cord blood transplantation on days 0-1. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 7 and continuing until blood counts recover.

Patients are followed monthly for 6 months; at 9, 12, 14, 16, 18, and 24 months; and then annually thereafter.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically confirmed diagnoses:

  * Acquired severe aplastic anemia

    * Meets at least 2 of the following criteria:

      * Granulocyte count less than 500/mm^3
      * Platelet count less than 20,000/mm^3
      * Absolute reticulocyte count less than 20,000/mm^3 (after correction for hematocrit)
    * Unresponsive to OR recurrent disease after prior treatment with anti-thymocyte globulin and/or cyclosporine
  * Acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * Failed induction therapy
    * In first complete remission (CR) with any of the following high-risk features:

      * Stem cell or biphenotype classification (M0)
      * Erythroleukemia (M6)
      * Acute megakaryocytic leukemia (M7)
      * Cytogenetic markers indicative of poor prognosis
      * t(15;17) translocation and failed first-line induction therapy OR there is molecular evidence of persistent disease
      * t(8;21) and inv(16) translocations and failed first-line induction therapy
    * In early relapse*
    * In second or subsequent remission
    * Recurrent disease after prior autologous stem cell transplantation (SCT) NOTE: *No refractory relapse
  * Acute lymphoblastic leukemia, meeting 1 of the following criteria:

    * In early relapse*
    * In second or subsequent remission
    * In first CR with the following high-risk features:

      * t(4;11) or t(9;22) translocation
      * Hyperleukocytosis (initial WBC greater than 30,000/mm^3)
      * Failed to achieve CR by day 28 of standard induction therapy
    * Recurrent disease after prior autologous SCT NOTE: *No refractory relapse
  * Chronic myelogenous leukemia

    * Chronic or accelerated phase that has failed medical management
    * Blastic phase allowed after reinduction chemotherapy induces chronic phase
  * Myelodysplastic syndromes meeting 1 of the following criteria:

    * Refractory to medical management
    * Presence of cytogenetic abnormalities predictive of transformation to acute leukemia, including the following:

= 5q- = 7q-

* Monosomy 7 and trisomy 8
* Evidence of evolution to AML (e.g., refractory anemia with excess blasts [RAEB], or RAEB in transformation)

  * Chronic lymphocytic leukemia

    * Refractory to treatment including fludarabine-based therapy
    * Recurrent disease after prior autologous SCT
  * Multiple myeloma

    * Recurrent disease after prior autologous SCT
    * Beyond first CR or failed induction therapy
    * Disease is sensitive to pretransplantation cytoreduction
  * Hodgkin's lymphoma

    * Beyond first CR or failed induction therapy
    * Disease is sensitive to pretransplantation cytoreduction
  * Non-Hodgkin's lymphoma (NHL)

    * Recurrent disease after prior autologous SCT
    * Beyond first CR or failed induction therapy
    * Disease is sensitive to pretransplantation cytoreduction
    * Mantle zone NHL allowed after induction therapy
  * Myeloproliferative disorders

    * Refractory to medical management
    * Allografting required unless grade 3 or greater myelofibrosis by bone marrow biopsy

      * No HLA-matched sibling donor available
      * Ineligible for a myeloablative conditioning regimen due to advanced age (over 55), extensive prior therapy, and/or other comorbidities
      * If under age 55, must meet at least 1 of the following criteria:
  * Received extensive prior therapy
  * Organ toxicity or infection precluding eligibility for allogeneic transplantation with full ablation conditioning

    * Availability of 2-5 umbilical cord blood units that are at least a 4/6 HLA match
    * No active CNS disease
    * No primary or grade 3 or 4 myelofibrosis

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Karnofsky 70-100% (for patients 16 years of age and older)
* Lansky 50-100% (for patients under 16 years of age)

Life expectancy

* At least 3 months

Hematopoietic

* See Disease Characteristics

Hepatic

* ALT/AST less than 4 times normal
* Bilirubin less than 2.0 mg/dL (unless due to hepatic infiltration by primary malignancy)

Renal

* Creatinine clearance greater than 40 mL/min

Cardiovascular

* Shortening fraction or ejection fraction greater than 40% of normal value for age by echocardiogram or radionuclide scan

Pulmonary

* FVC and FEV_1 greater than 60% of predicted
* DLCO greater than 60% of predicted (adult patients)
* Clearance by pulmonologist required if patient cannot perform pulmonary function tests

Other

* Not pregnant or nursing
* No uncontrolled active infection (viral, bacterial, or fungal)
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 3 months since prior autologous stem cell transplantation

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from prior therapy
* No other concurrent investigational agents that would preclude study participation or increase risk to patient

  * Investigational diagnostic procedures allowed

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival by disease assessment | at 28 and 100 days and then at 6, 9, 12, 18, and 24 months

SECONDARY OUTCOMES:
Umbilical cord blood donor engraftment by chimerism and complete blood count (CBC) | monthly for 6 months and then at 9, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Cooper, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States